CLINICAL TRIAL: NCT04108104
Title: Double-blind, Randomised, Parallel-group, Three-arm, Dose Range, Placebo-controlled, Proof-of-concept Study to Evaluate the Efficacy, Tolerability and Safety of a Combination of Cypropheptadine and Prazosin on Alcohol Consumption in Patients With Severe Alcohol Use Disorder
Brief Title: Clinical Outcome of a Patented Pharmaceutical Composition (KT-110) to Treat Alcohol Use Disorder While Avoiding Major Side Effects
Acronym: COCKTAIL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kinnov Therapeutics (Other)
Collaborators: ECSOR (Unknown)
Responsible Party: Sponsor
Organization: Greenpharma S.A.S. (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KT-100-001
Record Dates: First submitted 2019-09-25; First posted 2019-09-27 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism | interventions — Cyproheptadine; Prazosin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low-dose group (Experimental): Periactine® (Cyproheptadine 8 mg/day; two times 4 mg: morning and evening) and Alpress® (5 mg once a day slow-release: evening administration).
  Interventions: Drug: Cyproheptadine; Drug: Alpress LP
- High-dose group (Experimental): Periactine® (Cyproheptadine 12 mg/day; three times 4 mg: morning, noon and evening) and Alpress® (10 mg [2 tablets of 5 mg] once a day slow-release: evening administration)
  Interventions: Drug: Cyproheptadine; Drug: Alpress LP
- Placebo group (Placebo Comparator): Placebo of Periactine® (three times per day: morning, noon and evening) and placebo of Alpress® (once a day: evening)
  Interventions: Drug: Cyproheptadine; Drug: Alpress LP

INTERVENTIONS:
Drug: Cyproheptadine — 3-month treatment
  Other Names: Periactine®
Drug: Alpress LP — 3-month treatment
  Other Names: Prazosin

SUMMARY:
Double-blind randomised, parallel-group, three-arm, multicentre, placebo-controlled study The primary objective is to demonstrate the superiority of the combination of Periactine® (cyproheptadine 8 mg/day or 12 mg/day) and Alpress® (prazosin 5 mg/day or 10 mg/day) over placebo on the reduction of the total alcohol consumption (TAC), in alcohol-dependent patients.

180 patients will be randomised into the two treatment groups (N=60 in the low-dose group and N=60 in the high-dose group) and the placebo group (N=60).

ELIGIBILITY:
Inclusion Criteria:

* Severe alcohol use disorder
* High-risk alcohol consumption

Exclusion Criteria:

* Patient with orthostatic hypotension
* Patient with hypotension
* History of uncontrolled hypertension
* Patient at risk for urinary retention associated with urethroprostatic disorders
* Patient with a clinically-active malignancy
* Patient with a confirmed cirrhosis
* History of bronchial asthma
* History of uncontrolled hyperthyroidism
* History of cardiovascular disease not under control
* Severe psychiatric disorder
* History of alcohol withdrawal syndrome

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2019-11-30 (Actual); Primary Completion 2021-10-28 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Change in the mean quantity of alcohol consumed per day in the three groups | weeks 9 to 12

CONTACTS AND LOCATIONS:
Overall Officials: Alain Puech, Study Director — Kinnov Therapeutics
Locations (35):
- France (35):
  - Centre Hospitalier d'Abbeville, Abbeville
  - Centre d'Addictologie "Pierre-Fouquet" - CHD La Candélie, Agen
  - clinique de la Bréhonnière, Astillé
  - Centre de Soins, d'Accompagnement et de Prévention en addictologie Bizia, Bayonne
  - Centre Hospitalier de la Côte Basque - Service d'addictologie, Bayonne
  - Cabinet Médical, Bersée
  - CHRU Brest - Hôpital Cavale Blanche, Brest
  - HIA Clermont Tonnerre, Brest
  - Service Universitaire d'Addictologie de Lyon - Centre Hospitalier Le Vinatier, Bron
  - Centre Hospitalier Universitaire de Clermont-Ferrand, Clermont-Ferrand
  - Centre Hospitalier Intercommunal de Créteil - Service Hépato-Gastro-entérologie, Créteil
  - Centre Hospitalier Universitaire de Dijon - Service d'addictologie, Dijon
  - Centre Hospitalier Annecy Genevois, Épagny
  - Centre Hospitalier Camille Claudel, La Couronne
  - Centre Hospitalier de La Rochelle, La Rochelle
  - Centre Hospitalier Emile-Roux, Le Puy-en-Velay
  - Centre hospitalier Esquirol - Pôle d'addictologie en Limousin, Limoges
  - Centre Hospitalier Universitaire de Lyon - Hôpital de la Croix Rousse, Lyon
  - CHU Provences-Alpes Côte d'Azur Hôpital Publique, Marseille
  - Clinique Saint Barnabé, Marseille
  - Centre Hospitalier Régional Universitaire Saint Eloi - Service d'addictologie et complications somatiques, Montpellier
  - Hôpital St-Julien, Nancy
  - Centre Hospitalier Universitaire de Nantes - site Hôtel-Dieu, Nantes
  - Centre Hospitalier universitaire de Nice - Hôpital Archet II, Nice
  - Hôpital Universitaire Carémeau, Nîmes
  - Centre Hospitalier Régional d'Orléans - Hôpital La Source - Service d'hépato-gastro-entérologie et oncologie digestive, Orléans
  - Centre Médico-Psychologique Saint-Marc, Orléans
  - Centre Hospitalier Sainte-Anne, Paris
  - Hôpital Fernand-Widal, Paris
  - Centre Hospitalier de Pau - Unité d'addictologie, Pau
  - Centre Hospitalier Universitaire de Rennes - Hôpital Pontchaillou - Centre hépato-digestif, Rennes
  - Centre Ambulatoire de Santé Mentale, Saint-Martin-d'Hères
  - Centre Hospitalier de Saint-Nazaire, Saint-Nazaire
  - Association Hospitalière de Bourgogne Franche-Comté, Saint-Rémy
  - cabinet médical du Dr El-Ayoubi, Tours

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Aubin HJ, Berlin I, Guiraud J, Bruhwyler J, Batel P, Perney P, Trojak B, Bendimerad P, Guillou M, Bisch M, Grall-Bronnec M, Labarriere D, Delsart D, Questel F, Moirand R, Bernard P, Trovero F, Pham HP, Tassin JP, Puech A. Prazosin and cyproheptadine in combination in the treatment of alcohol use disorder: A randomized, double-blind, placebo-controlled trial. Addiction. 2024 Jul;119(7):1211-1223. doi: 10.1111/add.16484. Epub 2024 Apr 10. PMID 38597214